CLINICAL TRIAL: NCT04666441
Title: A Phase 2 Study to Assess the Virologic Efficacy of REGN10933+REGN10987 Across Different Dose Regimens in Outpatients With SARS-CoV-2 Infection
Brief Title: COVID-19 Study Assessing the Virologic Efficacy of REGN10933+REGN10987 Across Different Dose Regimens in Adult Outpatients With SARS-CoV-2 Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R10933-10987-COV-20145
Record Dates: First submitted 2020-12-10; First posted 2020-12-14 (Actual); Results first posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: COVID-19
Keywords: Coronavirus disease 2019 (COVID-19); Severe acute respiratory syndrome coronavirus 2 (SARS-COV-2) coronavirus; Non-hospitalized
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — casirivimab and imdevimab drug combination; casirivimab; imdevimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- IV Dose 1 (Experimental): Combination therapy intravenous (IV) single dose
  Interventions: Drug: REGN10933+REGN10987 combination therapy
- IV Dose 2 (Experimental): Combination therapy IV single dose
  Interventions: Drug: REGN10933+REGN10987 combination therapy
- IV Dose 3 (Experimental): Combination therapy IV single dose
  Interventions: Drug: REGN10933+REGN10987 combination therapy
- IV Dose 4 (Experimental): Combination therapy IV single dose
  Interventions: Drug: REGN10933+REGN10987 combination therapy
- Placebo IV Dose (Experimental): Matching placebo IV single dose
  Interventions: Drug: Placebo
- SC Dose 1 (Experimental): Combination therapy subcutaneous (SC) single dose
  Interventions: Drug: REGN10933+REGN10987 combination therapy
- SC Dose 2 (Experimental): Combination therapy SC single dose
  Interventions: Drug: REGN10933+REGN10987 combination therapy
- Placebo SC Dose (Experimental): Matching placebo SC single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: REGN10933+REGN10987 combination therapy — Administered IV or SC single dose
  Other Names: REGN-COV2; REGEN-COV™; Ronapreve™; casirivimab; imdevimab
  Arms: IV Dose 1; IV Dose 2; IV Dose 3; IV Dose 4; SC Dose 1; SC Dose 2
Drug: Placebo — Administered IV or SC single dose to match
  Arms: Placebo IV Dose; Placebo SC Dose

SUMMARY:
The primary objective of the study is to assess the virologic efficacy of REGN10933+REGN10987 across different intravenous and subcutaneous doses compared to placebo.

The secondary objectives of the study are:

* To evaluate additional indicators of virologic efficacy of REGN10933+REGN10987 compared to placebo
* To evaluate the safety and tolerability of REGN10933+REGN10987 compared to placebo
* To assess the concentrations of REGN10933 and REGN10987 in serum over time
* To assess the immunogenicity of REGN10933 and REGN10987

ELIGIBILITY:
Key Inclusion Criteria:

* Has SARS-CoV-2-positive diagnostic test from a sample collected ≤72 hours prior to randomization, as defined by the protocol
* Low-risk symptomatic patient: Has symptoms consistent with COVID-19 (as determined by the investigator) with onset ≤7 days before randomization, and meets all of the following 8 criteria:

  1. Age ≤50
  2. No obesity, with obesity defined as BMI ≥30 kg/m2
  3. Does not have cardiovascular disease or hypertension
  4. Does not have chronic lung disease or asthma
  5. Does not have type 1 or type 2 diabetes mellitus
  6. Does not have chronic kidney disease, with or without dialysis
  7. Does not have chronic liver disease
  8. Is not pregnant or
* Asymptomatic patient: Has had no symptoms consistent with COVID-19 (as determined by the investigator) occurring at any time <2 months prior to randomization
* Maintains O2 saturation ≥93% on room air

Key Exclusion Criteria:

* Was admitted to a hospital for COVID-19 prior to randomization, or is hospitalized (inpatient) for any reason at randomization
* Has a known positive SARS-CoV-2 serologic test
* Has a positive SARS-CoV-2 antigen or molecular diagnostic test from a sample collected >72 hours prior to randomization
* Is immunosuppressed, based on investigator's assessment
* Has participated, or is participating, in a clinical research study evaluating COVID-19 convalescent plasma, mAbs against SARS-CoV-2, or intravenous immunoglobulin (IVIG) within 3 months or within 5 half-lives of the investigational product (whichever is longer) prior to the screening visit
* Prior, current, or planned future use of any of the following treatments: COVID-19 convalescent plasma, mAbs against SARS-CoV-2, (eg, bamlanivimab), IVIG (any indication), systemic corticosteroids (any indication), or COVID-19 treatments (authorized, approved, or investigational)
* Prior use (prior to randomization), current use (at randomization), or planned use (within time period given per CDC guidance but no sooner than 22 days of study drug administration) of any authorized or approved vaccine for COVID-19
* Has known active infection with influenza or other non-SARS-CoV-2 respiratory pathogen, confirmed by a diagnostic test
* Has participated, is participating, or plans to participate in a clinical research study evaluating any authorized, approved, or investigational vaccine for COVID-19

NOTE: Other protocol defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1149 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2021-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (51):
- United States (51):
  - Regeneron Study Site, Mesa, Arizona
  - Regeneron Study Site, Tucson, Arizona
  - Regeneron Study Site, Canoga Park, California
  - Regeneron Study Site, Long Beach, California
  - Regeneron Study Site, Los Angeles, California
  - Regeneron Study Site, Rolling Hills Estates, California
  - Regeneron Study Site, San Francisco, California
  - Regeneron Study Site, Santa Monica, California
  - Regeneron Study Site, Stanford, California
  - Regeneron Study Site, Colorado Springs, Colorado
  - Regeneron Study Site, Washington D.C., District of Columbia
  - Regeneron Study Site, DeLand, Florida
  - Regeneron Study Site, Ft. Pierce, Florida
  - Regeneron Study Site, Hialeah, Florida
  - Regeneron Study Site, Maitland, Florida
  - Regeneron Study Site, Miami, Florida
  - Regeneron Study Site, St. Petersburg, Florida
  - Regeneron Study Site, Tampa, Florida
  - Regeneron Study Site, West Palm Beach, Florida
  - Regeneron Study Site, Winter Haven, Florida
  - Regeneron Study Site, Winter Park, Florida
  - Regeneron Study Site, Atlanta, Georgia
  - Regeneron Study Site, Columbus, Georgia
  - Regeneron Study Site, Downers Grove, Illinois
  - Regeneron Study Site, Ames, Iowa
  - Regeneron Study Site, Iowa City, Iowa
  - Regeneron Study Site, Lake Charles, Louisiana
  - Regeneron Study Site, Marrero, Louisiana
  - Regeneron Study Site, Shreveport, Louisiana
  - Regeneron Study Site, Baltimore, Maryland
  - Regeneron Study Site, Las Vegas, Nevada
  - Regeneron Study Site, Teaneck, New Jersey
  - Regeneron Study Site, New York, New York
  - Regeneron Study Site, The Bronx, New York
  - Regeneron Study Site, Charlotte, North Carolina
  - Regeneron Study Site, Durham, North Carolina
  - Regeneron Study Site, Wilmington, North Carolina
  - Regeneron Study Site, Columbus, Ohio
  - Regeneron Study Site, Dayton, Ohio
  - Regeneron Study Site, Philadelphia, Pennsylvania
  - Regeneron Study Site, Charleston, South Carolina
  - Regeneron Study Site, Clinton, South Carolina
  - Regeneron Study Site, Amarillo, Texas
  - Regeneron Study Site, Corpus Christi, Texas
  - Regeneron Study Site, Houston, Texas
  - Regeneron Study Site, Pearland, Texas
  - Regeneron Study Site, Red Oak, Texas
  - Regeneron Study Site, San Antonio, Texas
  - Regeneron Study Site, Splendora, Texas
  - Regeneron Study Site, Tyler, Texas
  - Regeneron Study Site, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

REFERENCES:
- [Derived] Portal-Celhay C, Forleo-Neto E, Eagan W, Musser BJ, Davis JD, Turner KC, Norton T, Hooper AT, Hamilton JD, Pan C, Mahmood A, Baum A, Kyratsous CA, Kim Y, Parrino J, Kampman W, Roque-Guerrero L, Stoici R, Fatakia A, Soo Y, Geba GP, Kowal B, DiCioccio AT, Stahl N, Lipsich L, Braunstein N, Herman GA, Yancopoulos GD, Weinreich DM; COVID-19 Phase 2 Dose-Ranging Study Team. Virologic Efficacy of Casirivimab and Imdevimab COVID-19 Antibody Combination in Outpatients With SARS-CoV-2 Infection: A Phase 2 Dose-Ranging Randomized Clinical Trial. JAMA Netw Open. 2022 Aug 1;5(8):e2225411. doi: 10.1001/jamanetworkopen.2022.25411. PMID 35969402
- [Derived] Hirsch C, Park YS, Piechotta V, Chai KL, Estcourt LJ, Monsef I, Salomon S, Wood EM, So-Osman C, McQuilten Z, Spinner CD, Malin JJ, Stegemann M, Skoetz N, Kreuzberger N. SARS-CoV-2-neutralising monoclonal antibodies to prevent COVID-19. Cochrane Database Syst Rev. 2022 Jun 17;6(6):CD014945. doi: 10.1002/14651858.CD014945.pub2. PMID 35713300
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1186 participants were screened and 1149 participants randomized and treated. Reasons for discontinuation at screening phase: 26-Screen Failure, 8-Subject Decision, 1-Sponsor Request, 1-Other. 1 randomized participant was not treated due to lack of supplies.
Groups:
- Placebo IV Dose: Participants received a single intravenous dose of placebo matching REGN10933+REGN10987
- 300mg IV: Participants received a single 300mg intravenous dose of REGN10933+REGN10987
- 600mg IV: Participants received a single 600mg intravenous dose of REGN10933+REGN10987
- 1200mg IV: Participants received a single 1200mg intravenous dose of REGN10933+REGN10987
- 2400mg IV: Participants received a single 2400mg intravenous dose of REGN10933+REGN10987
- Placebo SC Dose: Participants received a single subcutaneous dose of placebo matching REGN10933+REGN10987
- 600mg SC: Participants received a single 600mg subcutaneous dose of REGN10933+REGN10987
- 1200mg SC: Participants received a single 1200mg subcutaneous dose of REGN10933+REGN10987
Period: Overall Study
Arm/Group | Placebo IV Dose | 300mg IV | 600mg IV | 1200mg IV | 2400mg IV | Placebo SC Dose | 600mg SC | 1200mg SC
Started (Started = Randomized and treated) | 82 | 165 | 162 | 165 | 166 | 82 | 163 | 164
Completed | 80 | 160 | 158 | 161 | 166 | 79 | 158 | 160
Not Completed | 2 | 5 | 4 | 4 | 0 | 3 | 5 | 4
Not completed — Lost to Follow-up | 1 | 4 | 1 | 3 | 0 | 2 | 2 | 2
Not completed — Subject Decision | 1 | 1 | 3 | 1 | 0 | 1 | 3 | 2

BASELINE CHARACTERISTICS:
Population: Randomized participants who received any study drug; based on the treatment received (as treated)
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo IV Dose | 300mg IV | 600mg IV | 1200mg IV | 2400mg IV | Placebo SC Dose | 600mg SC | 1200mg SC | Total
Number analyzed (Participants) | 82 | 165 | 162 | 165 | 166 | 82 | 163 | 164 | 1149
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.5 (10.15) | 33.9 (8.99) | 34.2 (10.08) | 34.4 (9.81) | 33.9 (9.24) | 36.3 (9.88) | 33.5 (9.50) | 33.0 (10.18) | 34.0 (9.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 87 | 73 | 92 | 91 | 39 | 82 | 85 | 600
  Male | 31 | 78 | 89 | 73 | 75 | 43 | 81 | 79 | 549
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 67 | 58 | 60 | 73 | 32 | 68 | 62 | 446
  Not Hispanic or Latino | 55 | 96 | 98 | 102 | 91 | 49 | 94 | 99 | 684
  Unknown or Not Reported | 1 | 2 | 6 | 3 | 2 | 1 | 1 | 3 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 5
  Asian | 11 | 6 | 7 | 12 | 3 | 4 | 12 | 12 | 67
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 3
  Black or African American | 3 | 11 | 8 | 13 | 17 | 2 | 7 | 11 | 72
  White | 66 | 141 | 138 | 131 | 141 | 72 | 141 | 136 | 966
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 5 | 6 | 7 | 5 | 4 | 2 | 5 | 36
Viral Load in Nasopharyngeal Swab Samples [Mean (Standard Deviation); unit: log10 copies/mL] — Population: Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) results from central lab
  log10 copies/mL
    number analyzed (Participants) | 80 | 162 | 161 | 164 | 164 | 81 | 162 | 164 | 1138
    (all) | 5.98 (2.753) | 6.20 (2.697) | 5.70 (3.171) | 5.87 (2.656) | 6.12 (2.521) | 6.28 (2.521) | 6.15 (2.481) | 5.90 (2.832) | 6.01 (2.719)

OUTCOME MEASURES:

1. Primary Outcome: Time-Weighted Average Daily Change From Day 1 in Viral Load in NP Swab Samples
Description: Time-weighted average daily change from Day 1 in viral load (log10 copies/mL), as measured by reverse transcription quantitative polymerase chain reaction (RT-qPCR) in nasopharyngeal (NP) swab samples.
Time Frame: Day 1 to Day 7
Population: Seronegative modified Full Analysis Set (Seronegative mFAS): Participants in the Full Analysis Set (Overall mFAS) who were seronegative at baseline
Measure: Least Squares Mean (Standard Error); unit: log10 copies/mL
Groups:
- Pooled Placebo (IV + SC): Participants received a single intravenous dose of placebo matching REGN10933+REGN10987 or a single subcutaneous dose of placebo matching REGN10933+REGN10987
Arm/Group | Pooled Placebo (IV + SC) | 300mg IV | 600mg IV | 1200mg IV | 2400mg IV | 600mg SC | 1200mg SC
Number analyzed (Participants) | 74 | 76 | 66 | 67 | 61 | 71 | 71
log10 copies/mL | -1.68 (0.11) | -2.25 (0.11) | -2.34 (0.12) | -2.24 (0.12) | -2.40 (0.12) | -2.24 (0.12) | -2.24 (0.12)
Statistical Analysis 1: Comparison: Pooled Placebo (IV + SC) vs 300mg IV; Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p = 0.0004, ANCOVA; Difference of LS Means = -0.57, 95% CI 2-sided [-0.88 to -0.25], Standard Error of Mean 0.16
Statistical Analysis 2: Comparison: Pooled Placebo (IV + SC) vs 600mg IV; Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.66, 95% CI 2-sided [-0.99 to -0.34], Standard Error of Mean 0.17
Statistical Analysis 3: Comparison: Pooled Placebo (IV + SC) vs 1200mg IV; Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p = 0.0007, ANCOVA; Difference of LS Means = -0.56, 95% CI 2-sided [-0.89 to -0.24], Standard Error of Mean 0.16
Statistical Analysis 4: Comparison: Pooled Placebo (IV + SC) vs 2400mg IV; Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.71, 95% CI 2-sided [-1.05 to -0.38], Standard Error of Mean 0.17
Statistical Analysis 5: Comparison: Pooled Placebo (IV + SC) vs 600mg SC; Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p = 0.0006, ANCOVA; Difference of LS Means = -0.56, 95% CI [-0.88 to -0.24], Standard Error of Mean 0.16
Statistical Analysis 6: Comparison: Pooled Placebo (IV + SC) vs 1200mg SC; Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p = 0.0007, ANCOVA; Difference of LS Means = -0.56, 95% CI [-0.87 to -0.24], Standard Error of Mean 0.16

2. Secondary Outcome: Time-Weighted Average Daily Change From Day 1 in Viral Load
Description: Time-weighted average daily change from Day 1 in viral load (log10 copies/mL) as measured by reverse transcription quantitative polymerase chain reaction (RT-qPCR) in nasopharyngeal (NP) swab samples.
Time Frame: Day 1 to Day 5
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: log10 copies/mL
Arm/Group | Pooled Placebo (IV + SC) | 300mg IV | 600mg IV | 1200mg IV | 2400mg IV | 600mg SC | 1200mg SC
Number analyzed (Participants) | 105 | 104 | 96 | 94 | 90 | 99 | 107
log10 copies/mL | -1.19 (0.09) | -1.66 (0.09) | -1.76 (0.09) | -1.77 (0.09) | -1.68 (0.10) | -1.56 (0.09) | -1.61 (0.09)
Statistical Analysis 1: Comparison: Pooled Placebo (IV + SC) vs 300mg IV; Test type: Superiority; p = 0.0002, ANCOVA; Difference of LS Means = -0.47, 95% CI [-0.72 to -0.23], Standard Error of Mean 0.13
Statistical Analysis 2: Comparison: Pooled Placebo (IV + SC) vs 600mg IV; Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.57, 95% CI [-0.82 to -0.32], Standard Error of Mean 0.13
Statistical Analysis 3: Comparison: Pooled Placebo (IV + SC) vs 1200mg IV; Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.58, 95% CI [-0.83 to -0.33], Standard Error of Mean 0.13
Statistical Analysis 4: Comparison: Pooled Placebo (IV + SC) vs 2400mg IV; Test type: Superiority; p = 0.0002, ANCOVA; Difference of LS Means = -0.49, 95% CI [-0.75 to -0.24], Standard Error of Mean 0.13
Statistical Analysis 5: Comparison: Pooled Placebo (IV + SC) vs 600mg SC; Test type: Superiority; p = 0.0040, ANCOVA; Difference of LS Means = -0.37, 95% CI [-0.62 to -0.12], Standard Error of Mean 0.13
Statistical Analysis 6: Comparison: Pooled Placebo (IV + SC) vs 1200mg SC; Test type: Superiority; p = 0.0007, ANCOVA; Difference of LS Means = -0.42, 95% CI [-0.67 to -0.18], Standard Error of Mean 0.12

3. Secondary Outcome: Time-Weighted Average Daily Change From Day 1 in Viral Load in Participants With High Viral Load at Baseline
Description: Time-weighted average daily change from Day 1 in viral load (log10 copies/mL) as measured by reverse transcription quantitative polymerase chain reaction (RT-qPCR) in nasopharyngeal (NP) swab samples. in any participant with a viral load greater than 10,000 copies/mL at baseline.
Time Frame: Day 1 to Day 7
Population: Overall modified Full Analysis Set (Overall mFAS): All randomized participants with a positive central-lab determined SARS-CoV-2 RT-qPCR result from NP swab samples at randomization; based on the treatment received (as treated)
Measure: Least Squares Mean (Standard Error); unit: log10 copies/mL
Arm/Group | Pooled Placebo (IV + SC) | 300mg IV | 600mg IV | 1200mg IV | 2400mg IV | 600mg SC | 1200mg SC
Number analyzed (Participants) | 134 | 136 | 119 | 128 | 136 | 133 | 130
log10 copies/mL
  Baseline Viral Load is >10^4 copies/mL: number analyzed (Participants) | 131 | 132 | 118 | 124 | 133 | 131 | 126
  Baseline Viral Load is >10^4 copies/mL | -1.79 (0.09) | -2.36 (0.09) | -2.37 (0.09) | -2.41 (0.09) | -2.34 (0.09) | -2.30 (0.09) | -2.27 (0.09)
  Baseline Viral Load is >10^5 copies/mL: number analyzed (Participants) | 124 | 117 | 105 | 109 | 111 | 116 | 110
  Baseline Viral Load is >10^5 copies/mL | -1.82 (0.09) | -2.47 (0.09) | -2.51 (0.10) | -2.49 (0.09) | -2.46 (0.09) | -2.40 (0.09) | -2.38 (0.09)
  Baseline Viral Load is >10^6 copies/mL: number analyzed (Participants) | 102 | 97 | 97 | 95 | 94 | 97 | 97
  Baseline Viral Load is >10^6 copies/mL | -1.92 (0.10) | -2.62 (0.10) | -2.63 (0.10) | -2.64 (0.10) | -2.62 (0.10) | -2.47 (0.10) | -2.52 (0.10)
  Baseline Viral Load is >10^7 copies/mL: number analyzed (Participants) | 66 | 76 | 75 | 62 | 69 | 71 | 66
  Baseline Viral Load is >10^7 copies/mL | -1.89 (0.11) | -2.77 (0.11) | -2.83 (0.11) | -2.82 (0.12) | -2.72 (0.11) | -2.52 (0.11) | -2.73 (0.11)
Statistical Analysis 1: Comparison: Pooled Placebo (IV + SC) vs 300mg IV; Baseline Viral Load >10^4 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.57, 95% CI 2-sided [-0.82 to -0.33], Standard Error of Mean 0.13
Statistical Analysis 2: Comparison: Pooled Placebo (IV + SC) vs 300mg IV; Baseline Viral Load >10^5 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.65, 95% CI 2-sided [-0.90 to -0.40], Standard Error of Mean 0.13
Statistical Analysis 3: Comparison: Pooled Placebo (IV + SC) vs 300mg IV; Baseline Viral Load >10^6 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.70, 95% CI 2-sided [-0.97 to -0.42], Standard Error of Mean 0.14
Statistical Analysis 4: Comparison: Pooled Placebo (IV + SC) vs 300mg IV; Baseline Viral Load >10^7 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.88, 95% CI 2-sided [-1.19 to -0.58], Standard Error of Mean 0.16
Statistical Analysis 5: Comparison: Pooled Placebo (IV + SC) vs 600mg IV; Baseline Viral Load >10^4 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.58, 95% CI 2-sided [-0.84 to -0.33], Standard Error of Mean 0.13
Statistical Analysis 6: Comparison: Pooled Placebo (IV + SC) vs 600mg IV; Baseline Viral Load >10^5 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.69, 95% CI 2-sided [-0.95 to -0.43], Standard Error of Mean 0.13
Statistical Analysis 7: Comparison: Pooled Placebo (IV + SC) vs 600mg IV; Baseline Viral Load >10^6 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.71, 95% CI 2-sided [-0.98 to -0.44], Standard Error of Mean 0.14
Statistical Analysis 8: Comparison: Pooled Placebo (IV + SC) vs 600mg IV; Baseline Viral Load >10^7 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.95, 95% CI 2-sided [-1.25 to -0.64], Standard Error of Mean 0.16
Statistical Analysis 9: Comparison: Pooled Placebo (IV + SC) vs 1200mg IV; Baseline Viral Load >10^4 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.62, 95% CI 2-sided [-0.87 to -0.37], Standard Error of Mean 0.13
Statistical Analysis 10: Comparison: Pooled Placebo (IV + SC) vs 1200mg IV; Baseline Viral Load >10^5 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.67, 95% CI 2-sided [-0.93 to -0.42], Standard Error of Mean 0.13
Statistical Analysis 11: Comparison: Pooled Placebo (IV + SC) vs 1200mg IV; Baseline Viral Load >10^6 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.72, 95% CI 2-sided [-0.99 to -0.44], Standard Error of Mean 0.14
Statistical Analysis 12: Comparison: Pooled Placebo (IV + SC) vs 1200mg IV; Baseline Viral Load >10^7 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.93, 95% CI 2-sided [-1.25 to -0.61], Standard Error of Mean 0.16
Statistical Analysis 13: Comparison: Pooled Placebo (IV + SC) vs 2400mg IV; Baseline Viral Load >10^4 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.56, 95% CI 2-sided [-0.80 to -0.31], Standard Error of Mean 0.13
Statistical Analysis 14: Comparison: Pooled Placebo (IV + SC) vs 2400mg IV; Baseline Viral Load >10^5 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.64, 95% CI 2-sided [-0.89 to -0.38], Standard Error of Mean 0.13
Statistical Analysis 15: Comparison: Pooled Placebo (IV + SC) vs 2400mg IV; Baseline Viral Load >10^6 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.70, 95% CI 2-sided [-0.97 to -0.43], Standard Error of Mean 0.14
Statistical Analysis 16: Comparison: Pooled Placebo (IV + SC) vs 2400mg IV; Baseline Viral Load >10^7 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.84, 95% CI 2-sided [-1.15 to -0.52], Standard Error of Mean 0.16
Statistical Analysis 17: Comparison: Pooled Placebo (IV + SC) vs 600mg SC; Baseline Viral Load >10^4 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.51, 95% CI 2-sided [-0.76 to -0.27], Standard Error of Mean 0.13
Statistical Analysis 18: Comparison: Pooled Placebo (IV + SC) vs 600mg SC; Baseline Viral Load >10^5 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.58, 95% CI 2-sided [-0.83 to -0.33], Standard Error of Mean 0.13
Statistical Analysis 19: Comparison: Pooled Placebo (IV + SC) vs 600mg SC; Baseline Viral Load >10^6 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.55, 95% CI 2-sided [-0.82 to -0.28], Standard Error of Mean 0.14
Statistical Analysis 20: Comparison: Pooled Placebo (IV + SC) vs 600mg SC; Baseline Viral Load >10^7 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.63, 95% CI 2-sided [-0.95 to -0.32], Standard Error of Mean 0.16
Statistical Analysis 21: Comparison: Pooled Placebo (IV + SC) vs 1200mg SC; Baseline Viral Load >10^4 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p = 0.0002, ANCOVA; Difference of LS Means = -0.48, 95% CI 2-sided [-0.73 to -0.23], Standard Error of Mean 0.13
Statistical Analysis 22: Comparison: Pooled Placebo (IV + SC) vs 1200mg SC; Baseline Viral Load >10^5 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.56, 95% CI 2-sided [-0.82 to -0.31], Standard Error of Mean 0.13
Statistical Analysis 23: Comparison: Pooled Placebo (IV + SC) vs 1200mg SC; Baseline Viral Load >10^6 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.60, 95% CI 2-sided [-0.87 to -0.33], Standard Error of Mean 0.14
Statistical Analysis 24: Comparison: Pooled Placebo (IV + SC) vs 1200mg SC; Baseline Viral Load >10^7 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.84, 95% CI 2-sided [-1.16 to -0.52], Standard Error of Mean 0.16

4. Secondary Outcome: Time-Weighted Average Daily Change From Day 1 in Viral Load in Participants With High Viral Load at Baseline
Description: as for outcome 3
Time Frame: Day 1 to Day 5
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: log10 copies/mL
Arm/Group | Pooled Placebo (IV + SC) | 300mg IV | 600mg IV | 1200mg IV | 2400mg IV | 600mg SC | 1200mg SC
Number analyzed (Participants) | 128 | 131 | 115 | 124 | 132 | 128 | 126
log10 copies/mL
  Baseline Viral Load is >10^4 copies/mL | -1.28 (0.08) | -1.69 (0.08) | -1.73 (0.09) | -1.76 (0.09) | -1.68 (0.08) | -1.62 (0.08) | -1.61 (0.08)
  Baseline Viral Load is >10^5 copies/mL: number analyzed (Participants) | 121 | 116 | 102 | 109 | 109 | 114 | 109
  Baseline Viral Load is >10^5 copies/mL | -1.30 (0.08) | -1.77 (0.08) | -1.83 (0.09) | -1.81 (0.09) | -1.76 (0.09) | -1.69 (0.08) | -1.69 (0.09)
  Baseline Viral Load is >10^6 copies/mL: number analyzed (Participants) | 98 | 96 | 94 | 93 | 91 | 96 | 96
  Baseline Viral Load is >10^6 copies/mL | -1.38 (0.09) | -1.89 (0.09) | -1.92 (0.09) | -1.93 (0.09) | -1.91 (0.09) | -1.76 (0.09) | -1.79 (0.09)
  Baseline Viral Load is >10^7 copies/mL: number analyzed (Participants) | 62 | 76 | 72 | 61 | 67 | 69 | 66
  Baseline Viral Load is >10^7 copies/mL | -1.39 (0.11) | -1.99 (0.10) | -2.08 (0.10) | -2.08 (0.11) | -2.01 (0.10) | -1.76 (0.10) | -1.97 (0.10)
Statistical Analysis 1: Comparison: Pooled Placebo (IV + SC) vs 300mg IV; Baseline Viral Load >10^4 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p = 0.0005, ANCOVA; Difference of LS Means = -0.41, 95% CI 2-sided [-0.64 to -0.18], Standard Error of Mean 0.12
Statistical Analysis 2: Comparison: Pooled Placebo (IV + SC) vs 300mg IV; Baseline Viral Load >10^5 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.46, 95% CI 2-sided [-0.69 to -0.23], Standard Error of Mean 0.12
Statistical Analysis 3: Comparison: Pooled Placebo (IV + SC) vs 300mg IV; Baseline Viral Load >10^6 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.51, 95% CI 2-sided [-0.75 to -0.26], Standard Error of Mean 0.13
Statistical Analysis 4: Comparison: Pooled Placebo (IV + SC) vs 300mg IV; Baseline Viral Load >10^7 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.60, 95% CI 2-sided [-0.88 to -0.32], Standard Error of Mean 0.14
Statistical Analysis 5: Comparison: Pooled Placebo (IV + SC) vs 600mg IV; Baseline Viral Load >10^4 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p = 0.0003, ANCOVA; Difference of LS Means = -0.45, 95% CI 2-sided [-0.69 to -0.21], Standard Error of Mean 0.12
Statistical Analysis 6: Comparison: Pooled Placebo (IV + SC) vs 600mg IV; Baseline Viral Load >10^5 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.53, 95% CI 2-sided [-0.77 to -0.29], Standard Error of Mean 0.12
Statistical Analysis 7: Comparison: Pooled Placebo (IV + SC) vs 600mg IV; Baseline Viral Load >10^6 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.53, 95% CI 2-sided [-0.78 to -0.29], Standard Error of Mean 0.13
Statistical Analysis 8: Comparison: Pooled Placebo (IV + SC) vs 600mg IV; Baseline Viral Load >10^7 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.69, 95% CI 2-sided [-0.98 to -0.41], Standard Error of Mean 0.14
Statistical Analysis 9: Comparison: Pooled Placebo (IV + SC) vs 1200mg IV; Baseline Viral Load >10^4 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.48, 95% CI 2-sided [-0.72 to -0.25], Standard Error of Mean 0.12
Statistical Analysis 10: Comparison: Pooled Placebo (IV + SC) vs 1200mg IV; Baseline Viral Load >10^5 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.51, 95% CI 2-sided [-0.74 to -0.28], Standard Error of Mean 0.12
Statistical Analysis 11: Comparison: Pooled Placebo (IV + SC) vs 1200mg IV; Baseline Viral Load >10^6 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.54, 95% CI 2-sided [-0.79 to -0.30], Standard Error of Mean 0.13
Statistical Analysis 12: Comparison: Pooled Placebo (IV + SC) vs 1200mg IV; Baseline Viral Load >10^7 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.70, 95% CI 2-sided [-0.99 to -0.40], Standard Error of Mean 0.15
Statistical Analysis 13: Comparison: Pooled Placebo (IV + SC) vs 2400mg IV; Baseline Viral Load >10^4 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p = 0.0009, ANCOVA; Difference of LS Means = -0.39, 95% CI 2-sided [-0.63 to -0.16], Standard Error of Mean 0.12
Statistical Analysis 14: Comparison: Pooled Placebo (IV + SC) vs 2400mg IV; Baseline Viral Load >10^5 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p = 0.0001, ANCOVA; Difference of LS Means = -0.46, 95% CI 2-sided [-0.69 to -0.23], Standard Error of Mean 0.12
Statistical Analysis 15: Comparison: Pooled Placebo (IV + SC) vs 2400mg IV; Baseline Viral Load >10^6 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.52, 95% CI 2-sided [-0.77 to -0.27], Standard Error of Mean 0.13
Statistical Analysis 16: Comparison: Pooled Placebo (IV + SC) vs 2400mg IV; Baseline Viral Load >10^7 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p < 0.0001, ANCOVA; Difference of LS Means = -0.63, 95% CI 2-sided [-0.92 to -0.34], Standard Error of Mean 0.15
Statistical Analysis 17: Comparison: Pooled Placebo (IV + SC) vs 600mg SC; Baseline Viral Load >10^4 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p = 0.0046, ANCOVA; Difference of LS Means = -0.34, 95% CI 2-sided [-0.57 to -0.10], Standard Error of Mean 0.12
Statistical Analysis 18: Comparison: Pooled Placebo (IV + SC) vs 600mg SC; Baseline Viral Load >10^5 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p = 0.0011, ANCOVA; Difference of LS Means = -0.39, 95% CI 2-sided [-0.62 to -0.15], Standard Error of Mean 0.12
Statistical Analysis 19: Comparison: Pooled Placebo (IV + SC) vs 600mg SC; Baseline Viral Load >10^6 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p = 0.0029, ANCOVA; Difference of LS Means = -0.37, 95% CI 2-sided [-0.62 to -0.13], Standard Error of Mean 0.13
Statistical Analysis 20: Comparison: Pooled Placebo (IV + SC) vs 600mg SC; Baseline Viral Load >10^7 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p = 0.0120, ANCOVA; Difference of LS Means = -0.37, 95% CI 2-sided [-0.66 to -0.08], Standard Error of Mean 0.15
Statistical Analysis 21: Comparison: Pooled Placebo (IV + SC) vs 1200mg SC; Baseline Viral Load >10^4 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p = 0.0062, ANCOVA; Difference of LS Means = -0.33, 95% CI 2-sided [-0.56 to -0.09], Standard Error of Mean 0.12
Statistical Analysis 22: Comparison: Pooled Placebo (IV + SC) vs 1200mg SC; Baseline Viral Load >10^5 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p = 0.0011, ANCOVA; Difference of LS Means = -0.39, 95% CI 2-sided [-0.62 to -0.16], Standard Error of Mean 0.12
Statistical Analysis 23: Comparison: Pooled Placebo (IV + SC) vs 1200mg SC; Baseline Viral Load >10^6 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p = 0.0011, ANCOVA; Difference of LS Means = -0.41, 95% CI 2-sided [-0.66 to -0.17], Standard Error of Mean 0.13
Statistical Analysis 24: Comparison: Pooled Placebo (IV + SC) vs 1200mg SC; Baseline Viral Load >10^7 copies/mL Difference vs. Placebo (log10 copies/mL); Test type: Superiority; p = 0.0001, ANCOVA; Difference of LS Means = -0.58, 95% CI 2-sided [-0.87 to -0.29], Standard Error of Mean 0.15

5. Secondary Outcome: Number of Participants With High Viral Load
Description: Number of participants with viral load greater than 10,000 copies/mL, as measured by reverse transcription quantitative polymerase chain reaction (RT-qPCR) in nasopharyngeal (NP) swab samples.
Time Frame: Day 1, Day 3, Day 5, Day 7, Day 15, Day 22
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo (IV + SC) | 300mg IV | 600mg IV | 1200mg IV | 2400mg IV | 600mg SC | 1200mg SC
Number analyzed (Participants) | 109 | 108 | 100 | 97 | 93 | 103 | 111
Participants
  Day 1 Viral Load >10^4 copies/mL | 108 | 106 | 96 | 95 | 91 | 99 | 106
  Day 1 Viral Load >10^5 copies/mL | 104 | 99 | 92 | 89 | 84 | 93 | 95
  Day 1 Viral Load >10^6 copies/mL | 88 | 83 | 86 | 76 | 78 | 81 | 88
  Day 1 Viral Load >10^7 copies/mL | 60 | 67 | 64 | 54 | 58 | 63 | 62
  Day 3 Viral Load >10^4 copies/mL: number analyzed (Participants) | 106 | 107 | 97 | 94 | 92 | 102 | 106
  Day 3 Viral Load >10^4 copies/mL | 93 | 92 | 79 | 80 | 80 | 89 | 89
  Day 3 Viral Load >10^5 copies/mL: number analyzed (Participants) | 106 | 107 | 97 | 94 | 92 | 102 | 106
  Day 3 Viral Load >10^5 copies/mL | 83 | 68 | 63 | 67 | 61 | 68 | 75
  Day 3 Viral Load >10^6 copies/mL: number analyzed (Participants) | 106 | 107 | 97 | 94 | 92 | 102 | 106
  Day 3 Viral Load >10^6 copies/mL | 59 | 47 | 43 | 36 | 39 | 41 | 53
  Day 3 Viral Load >10^7 copies/mL: number analyzed (Participants) | 106 | 107 | 97 | 94 | 92 | 102 | 106
  Day 3 Viral Load >10^7 copies/mL | 29 | 15 | 15 | 14 | 14 | 25 | 23
  Day 5 Viral Load >10^4 copies/mL: number analyzed (Participants) | 105 | 104 | 96 | 94 | 90 | 99 | 107
  Day 5 Viral Load >10^4 copies/mL | 78 | 65 | 58 | 58 | 55 | 62 | 67
  Day 5 Viral Load >10^5 copies/mL: number analyzed (Participants) | 105 | 104 | 96 | 94 | 90 | 99 | 107
  Day 5 Viral Load >10^5 copies/mL | 53 | 31 | 20 | 30 | 29 | 29 | 31
  Day 5 Viral Load >10^6 copies/mL: number analyzed (Participants) | 105 | 104 | 96 | 94 | 90 | 99 | 107
  Day 5 Viral Load >10^6 copies/mL | 29 | 7 | 9 | 3 | 10 | 7 | 9
  Day 5 Viral Load >10^7 copies/mL: number analyzed (Participants) | 105 | 104 | 96 | 94 | 90 | 99 | 107
  Day 5 Viral Load >10^7 copies/mL | 14 | 0 | 3 | 0 | 0 | 5 | 2
  Day 7 Viral Load >10^4 copies/mL: number analyzed (Participants) | 107 | 106 | 99 | 93 | 92 | 102 | 107
  Day 7 Viral Load >10^4 copies/mL | 59 | 32 | 35 | 27 | 28 | 33 | 35
  Day 7 Viral Load >10^5 copies/mL: number analyzed (Participants) | 107 | 106 | 99 | 93 | 92 | 102 | 107
  Day 7 Viral Load >10^5 copies/mL | 32 | 9 | 9 | 7 | 13 | 9 | 9
  Day 7 Viral Load >10^6 copies/mL: number analyzed (Participants) | 107 | 106 | 99 | 93 | 92 | 102 | 107
  Day 7 Viral Load >10^6 copies/mL | 13 | 2 | 1 | 0 | 0 | 2 | 1
  Day 7 Viral Load >10^7 copies/mL: number analyzed (Participants) | 107 | 106 | 99 | 93 | 92 | 102 | 107
  Day 7 Viral Load >10^7 copies/mL | 5 | 1 | 0 | 0 | 0 | 0 | 1
  Day 15 Viral Load >10^4 copies/mL: number analyzed (Participants) | 106 | 104 | 98 | 92 | 92 | 100 | 107
  Day 15 Viral Load >10^4 copies/mL | 8 | 3 | 6 | 7 | 7 | 4 | 4
  Day 15 Viral Load >10^5 copies/mL: number analyzed (Participants) | 106 | 104 | 98 | 92 | 92 | 100 | 107
  Day 15 Viral Load >10^5 copies/mL | 4 | 1 | 2 | 3 | 1 | 1 | 0
  Day 15 Viral Load >10^6 copies/mL: number analyzed (Participants) | 106 | 104 | 98 | 92 | 92 | 100 | 107
  Day 15 Viral Load >10^6 copies/mL | 1 | 1 | 1 | 0 | 1 | 1 | 0
  Day 15 Viral Load >10^7 copies/mL: number analyzed (Participants) | 106 | 104 | 98 | 92 | 92 | 100 | 107
  Day 15 Viral Load >10^7 copies/mL | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Day 22 Viral Load >10^4 copies/mL: number analyzed (Participants) | 106 | 103 | 99 | 93 | 88 | 99 | 108
  Day 22 Viral Load >10^4 copies/mL | 3 | 0 | 3 | 0 | 4 | 1 | 3
  Day 22 Viral Load >10^5 copies/mL: number analyzed (Participants) | 106 | 103 | 99 | 93 | 88 | 99 | 108
  Day 22 Viral Load >10^5 copies/mL | 2 | 0 | 0 | 0 | 1 | 1 | 0
  Day 22 Viral Load >10^6 copies/mL: number analyzed (Participants) | 106 | 103 | 99 | 93 | 88 | 99 | 108
  Day 22 Viral Load >10^6 copies/mL | 1 | 0 | 0 | 0 | 1 | 0 | 0
  Day 22 Viral Load >10^7 copies/mL: number analyzed (Participants) | 106 | 103 | 99 | 93 | 88 | 99 | 108
  Day 22 Viral Load >10^7 copies/mL | 0 | 0 | 0 | 0 | 1 | 0 | 0

6. Secondary Outcome: Number of Participants With Viral Loads Below the Limit of Detection
Description: Number of participants with viral load less than 299 copies/mL, as measured by reverse transcription quantitative polymerase chain reaction (RT-qPCR) in nasopharyngeal (NP) swab samples.
Time Frame: Day 1, Day 3, Day 5, Day 7, Day 15, Day 22
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo (IV + SC) | 300mg IV | 600mg IV | 1200mg IV | 2400mg IV | 600mg SC | 1200mg SC
Number analyzed (Participants) | 109 | 108 | 100 | 97 | 93 | 103 | 111
Participants
  Day 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 3: number analyzed (Participants) | 106 | 107 | 97 | 94 | 92 | 102 | 106
  Day 3 | 3 | 1 | 4 | 3 | 1 | 1 | 5
  Day 5: number analyzed (Participants) | 105 | 104 | 96 | 94 | 90 | 99 | 107
  Day 5 | 6 | 11 | 10 | 12 | 12 | 11 | 12
  Day 7: number analyzed (Participants) | 107 | 106 | 99 | 93 | 92 | 102 | 107
  Day 7 | 19 | 22 | 16 | 14 | 18 | 25 | 19
  Day 15: number analyzed (Participants) | 106 | 104 | 98 | 92 | 92 | 100 | 107
  Day 15 | 55 | 68 | 58 | 54 | 50 | 67 | 65
  Day 22: number analyzed (Participants) | 106 | 103 | 99 | 93 | 88 | 99 | 108
  Day 22 | 73 | 78 | 74 | 70 | 62 | 81 | 84

7. Secondary Outcome: Number of Participants With Viral Loads Below the Lower Limit of Quantification
Description: Number of participants with viral load less than 714 copies/mL, as measured by reverse transcription quantitative polymerase chain reaction (RT-qPCR) in nasopharyngeal (NP) swab samples.
Time Frame: Day 1, Day 3, Day 5, Day 7, Day 15, Day 22
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo (IV + SC) | 300mg IV | 600mg IV | 1200mg IV | 2400mg IV | 600mg SC | 1200mg SC
Number analyzed (Participants) | 109 | 108 | 100 | 97 | 93 | 103 | 111
Participants
  Day 1 | 0 | 1 | 0 | 0 | 0 | 3 | 0
  Day 3: number analyzed (Participants) | 106 | 107 | 97 | 94 | 92 | 102 | 106
  Day 3 | 4 | 5 | 4 | 6 | 2 | 1 | 7
  Day 5: number analyzed (Participants) | 105 | 104 | 96 | 94 | 90 | 99 | 107
  Day 5 | 8 | 17 | 14 | 20 | 14 | 15 | 14
  Day 7: number analyzed (Participants) | 107 | 106 | 99 | 93 | 92 | 102 | 107
  Day 7 | 25 | 33 | 24 | 26 | 24 | 38 | 27
  Day 15: number analyzed (Participants) | 106 | 104 | 98 | 92 | 92 | 100 | 107
  Day 15 | 69 | 78 | 69 | 67 | 62 | 76 | 83
  Day 22: number analyzed (Participants) | 106 | 103 | 99 | 93 | 88 | 99 | 108
  Day 22 | 84 | 87 | 83 | 81 | 74 | 87 | 95

8. Secondary Outcome: Change From Day 1 in Viral Load as Measured by RT-qPCR in NP Swab Samples
Description: Change from Day 1 in Viral Load (log10 copies/mL) as Measured by Quantitative reverse transcription polymerase chain reaction (RT-qPCR) in nasopharyngeal (NP) Swab Samples
Time Frame: Day 3, Day 5, Day 7, Day 15, Day 22
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: log10 copies/mL
Arm/Group | Pooled Placebo (IV + SC) | 300mg IV | 600mg IV | 1200mg IV | 2400mg IV | 600mg SC | 1200mg SC
Number analyzed (Participants) | 109 | 108 | 100 | 97 | 93 | 103 | 111
log10 copies/mL
  Day 3 change from Day 1: number analyzed (Participants) | 106 | 107 | 97 | 94 | 92 | 102 | 106
  Day 3 change from Day 1 | -1.22 (0.13) | -1.71 (0.13) | -1.91 (0.14) | -1.85 (0.14) | -1.69 (0.14) | -1.55 (0.13) | -1.65 (0.13)
  Day 5 change from Day 1: number analyzed (Participants) | 105 | 104 | 96 | 94 | 90 | 99 | 107
  Day 5 change from Day 1 | -2.29 (0.16) | -3.24 (0.16) | -3.37 (0.16) | -3.32 (0.17) | -3.33 (0.17) | -3.19 (0.16) | -3.20 (0.16)
  Day 7 change from Day 1: number analyzed (Participants) | 107 | 106 | 99 | 93 | 92 | 102 | 107
  Day 7 change from Day 1 | -3.44 (0.16) | -4.24 (0.16) | -4.08 (0.16) | -4.10 (0.17) | -4.17 (0.17) | -4.33 (0.16) | -4.04 (0.16)
  Day 15 change from Day 1: number analyzed (Participants) | 106 | 104 | 98 | 92 | 92 | 100 | 107
  Day 15 change from Day 1 | -5.66 (0.16) | -6.11 (0.16) | -5.97 (0.17) | -5.91 (0.17) | -5.77 (0.17) | -6.17 (0.17) | -6.05 (0.16)
  Day 22 change from Day 1: number analyzed (Participants) | 106 | 103 | 99 | 93 | 88 | 99 | 108
  Day 22 change from Day 1 | -6.27 (0.13) | -6.58 (0.14) | -6.50 (0.14) | -6.56 (0.14) | -6.36 (0.15) | -6.69 (0.14) | -6.60 (0.13)
Statistical Analysis 1: Comparison: Pooled Placebo (IV + SC) vs 300mg IV; Difference vs. Placebo, by Day 3 (log10 copies/mL); Test type: Superiority; p = 0.0070, Mixed Model for Repeated Measures (MMRM); Difference of LS Means = -0.49, 95% CI [-0.85 to -0.14], Standard Error of Mean 0.18
Statistical Analysis 2: Comparison: Pooled Placebo (IV + SC) vs 600mg IV; Difference vs. Placebo, by Day 3 (log10 copies/mL); Test type: Superiority; p = 0.0002, Mixed Model for Repeated Measures (MMRM); Difference of LS Means = -0.69, 95% CI 2-sided [-1.06 to -0.33], Standard Error of Mean 0.19
Statistical Analysis 3: Comparison: Pooled Placebo (IV + SC) vs 1200mg IV; Difference vs. Placebo, by Day 3 (log10 copies/mL); Test type: Superiority; p = 0.0008, Mixed Model for Repeated Measures (MMRM); Difference of LS Means = -0.63, 95% CI [-1.00 to -0.26], Standard Error of Mean 0.19
Statistical Analysis 4: Comparison: Pooled Placebo (IV + SC) vs 2400mg IV; Difference vs. Placebo, by Day 3 (log10 copies/mL); Test type: Superiority; p = 0.0125, Mixed Model for Repeated Measures (MMRM); Difference of LS Means = -0.48, 95% CI [-0.85 to -0.10], Standard Error of Mean 0.19
Statistical Analysis 5: Comparison: Pooled Placebo (IV + SC) vs 600mg SC; Difference vs. Placebo, by Day 3 (log10 copies/mL); Test type: Superiority; p = 0.0696, Mixed Model for Repeated Measures (MMRM); Difference of LS Means = -0.34, 95% CI [-0.70 to 0.03], Standard Error of Mean 0.18
Statistical Analysis 6: Comparison: Pooled Placebo (IV + SC) vs 1200mg SC; Difference vs. Placebo, by Day 3 (log10 copies/mL); Test type: Superiority; p = 0.0187, Mixed Model for Repeated Measures (MMRM); Difference of LS Means = -0.43, 95% CI 2-sided [-0.79 to -0.07], Standard Error of Mean 0.18
Statistical Analysis 7: Comparison: Pooled Placebo (IV + SC) vs 300mg IV; Difference vs. Placebo, by Day 5 (log10 copies/mL); Test type: Superiority; p < 0.0001, Mixed Model for Repeated Measures (MMRM); Difference of LS Means = -0.96, 95% CI [-1.39 to -0.52], Standard Error of Mean 0.22
Statistical Analysis 8: Comparison: Pooled Placebo (IV + SC) vs 600mg IV; Difference vs. Placebo, by Day 5 (log10 copies/mL); Test type: Superiority; p < 0.0001, Mixed Model for Repeated Measures (MMRM); Difference of LS Means = -1.09, 95% CI [-1.53 to -0.64], Standard Error of Mean 0.23
Statistical Analysis 9: Comparison: Pooled Placebo (IV + SC) vs 1200mg IV; Difference vs. Placebo, by Day 5 (log10 copies/mL); Test type: Superiority; p < 0.0001, Mixed Model for Repeated Measures (MMRM); Difference of LS Means = -1.03, 95% CI [-1.48 to -0.59], Standard Error of Mean 0.23
Statistical Analysis 10: Comparison: Pooled Placebo (IV + SC) vs 2400mg IV; Difference vs. Placebo, by Day 5 (log10 copies/mL); Test type: Superiority; p < 0.0001, Mixed Model for Repeated Measures (MMRM); Difference of LS Means = -1.05, 95% CI [-1.50 to -0.60], Standard Error of Mean 0.23
Statistical Analysis 11: Comparison: Pooled Placebo (IV + SC) vs 600mg SC; Difference vs. Placebo, by Day 5 (log10 copies/mL); Test type: Superiority; p < 0.0001, Mixed Model for Repeated Measures (MMRM); Difference of LS Means = -0.90, 95% CI 2-sided [-1.34 to -0.46], Standard Error of Mean 0.22
Statistical Analysis 12: Comparison: Pooled Placebo (IV + SC) vs 1200mg SC; Difference vs. Placebo, by Day 5 (log10 copies/mL); Test type: Superiority; p < 0.0001, Mixed Model for Repeated Measures (MMRM); Difference of LS Means = -0.92, 95% CI [-1.35 to -0.48], Standard Error of Mean 0.22
Statistical Analysis 13: Comparison: Pooled Placebo (IV + SC) vs 300mg IV; Difference vs. Placebo, by Day 7 (log10 copies/mL); Test type: Superiority; p = 0.0004, Mixed Model for Repeated Measures (MMRM); Difference of LS Means = -0.79, 95% CI [-1.23 to -0.35], Standard Error of Mean 0.22
Statistical Analysis 14: Comparison: Pooled Placebo (IV + SC) vs 600mg IV; Difference vs. Placebo, by Day 7 (log10 copies/mL); Test type: Superiority; p = 0.0058, Mixed Model for Repeated Measures (MMRM); Difference of LS Means = -0.63, 95% CI [-1.08 to -0.18], Standard Error of Mean 0.23
Statistical Analysis 15: Comparison: Pooled Placebo (IV + SC) vs 1200mg IV; Difference vs. Placebo, by Day 7 (log10 copies/mL); Test type: Superiority; p = 0.0046, Mixed Model for Repeated Measures (MMRM); Difference of LS Means = -0.66, 95% CI [-1.11 to -0.20], Standard Error of Mean 0.23
Statistical Analysis 16: Comparison: Pooled Placebo (IV + SC) vs 2400mg IV; Difference vs. Placebo, by Day 7 (log10 copies/mL); Test type: Superiority; p = 0.0019, Mixed Model for Repeated Measures (MMRM); Difference of LS Means = -0.73, 95% CI [-1.18 to -0.27], Standard Error of Mean 0.23
Statistical Analysis 17: Comparison: Pooled Placebo (IV + SC) vs 600mg SC; Difference vs. Placebo, by Day 7 (log10 copies/mL); Test type: Superiority; p < 0.0001, Mixed Model for Repeated Measures (MMRM); Difference of LS Means = -0.89, 95% CI [-1.33 to -0.44], Standard Error of Mean 0.23
Statistical Analysis 18: Comparison: Pooled Placebo (IV + SC) vs 1200mg SC; Difference vs. Placebo, by Day 7 (log10 copies/mL); Test type: Superiority; p = 0.0079, Mixed Model for Repeated Measures (MMRM); Difference of LS Means = -0.60, 95% CI [-1.04 to -0.16], Standard Error of Mean 0.22
Statistical Analysis 19: Comparison: Pooled Placebo (IV + SC) vs 300mg IV; Difference vs. Placebo, by Day 15 (log10 copies/mL); Test type: Superiority; p = 0.0515, Mixed Model for Repeated Measures (MMRM); Difference of LS Means = -0.45, 95% CI [-0.90 to 0.00], Standard Error of Mean 0.23
Statistical Analysis 20: Comparison: Pooled Placebo (IV + SC) vs 600mg IV; Difference vs. Placebo, by Day 15 (log10 copies/mL); Test type: Superiority; p = 0.1864, Mixed Model for Repeated Measures (MMRM); Difference of LS Means = -0.31, 95% CI [-0.77 to 0.15], Standard Error of Mean 0.23
Statistical Analysis 21: Comparison: Pooled Placebo (IV + SC) vs 1200mg IV; Difference vs. Placebo, by Day 15 (log10 copies/mL); Test type: Superiority; p = 0.2866, Mixed Model for Repeated Measures (MMRM); Difference of LS Means = -0.25, 95% CI [-0.72 to 0.21], Standard Error of Mean 0.24
Statistical Analysis 22: Comparison: Pooled Placebo (IV + SC) vs 2400mg IV; Difference vs. Placebo, by Day 15 (log10 copies/mL); Test type: Superiority; p = 0.6470, Mixed Model for Repeated Measures (MMRM); Difference of LS Means = -0.11, 95% CI [-0.58 to 0.36], Standard Error of Mean 0.24
Statistical Analysis 23: Comparison: Pooled Placebo (IV + SC) vs 600mg SC; Difference vs. Placebo, by Day 15 (log10 copies/mL); Test type: Superiority; p = 0.0280, Mixed Model for Repeated Measures (MMRM); Difference of LS Means = -0.51, 95% CI [-0.97 to -0.06], Standard Error of Mean 0.23
Statistical Analysis 24: Comparison: Pooled Placebo (IV + SC) vs 1200mg SC; Difference vs. Placebo, by Day 15 (log10 copies/mL); Test type: Superiority; p = 0.0854, Mixed Models Analysis; Difference of LS Means = -0.39, 95% CI [-0.84 to 0.05], Standard Error of Mean 0.23
Statistical Analysis 25: Comparison: Pooled Placebo (IV + SC) vs 300mg IV; Difference vs. Placebo, by Day 22 (log10 copies/mL); Test type: Superiority; p = 0.1078, Mixed Model for Repeated Measures (MMRM); Difference of LS Means = -0.31, 95% CI 2-sided [-0.69 to 0.07], Standard Error of Mean 0.19
Statistical Analysis 26: Comparison: Pooled Placebo (IV + SC) vs 600mg IV; Difference vs. Placebo, by Day 22 (log10 copies/mL); Test type: Superiority; p = 0.2235, Mixed Model for Repeated Measures (MMRM); Difference of LS Means = -0.24, 95% CI [-0.62 to 0.14], Standard Error of Mean 0.19
Statistical Analysis 27: Comparison: Pooled Placebo (IV + SC) vs 1200mg IV; Difference vs. Placebo, by Day 22 (log10 copies/mL); Test type: Superiority; p = 0.1369, Mixed Model for Repeated Measures (MMRM); Difference of LS Means = -0.29, 95% CI [-0.68 to 0.09], Standard Error of Mean 0.20
Statistical Analysis 28: Comparison: Pooled Placebo (IV + SC) vs 2400mg IV; Difference vs. Placebo, by Day 22 (log10 copies/mL); Test type: Superiority; p = 0.6610, Mixed Model for Repeated Measures (MMRM); Difference of LS Means = -0.09, 95% CI [-0.48 to 0.31], Standard Error of Mean 0.20
Statistical Analysis 29: Comparison: Pooled Placebo (IV + SC) vs 600mg SC; Difference vs. Placebo, by Day 22 (log10 copies/mL); Test type: Superiority; p = 0.0284, Mixed Model for Repeated Measures (MMRM); Difference of LS Means = -0.43, 95% CI [-0.81 to -0.05], Standard Error of Mean 0.19
Statistical Analysis 30: Comparison: Pooled Placebo (IV + SC) vs 1200mg SC; Difference vs. Placebo, by Day 22 (log10 copies/mL); Test type: Superiority; p = 0.0800, Mixed Model for Repeated Measures (MMRM); Difference of LS Means = -0.33, 95% CI [-0.71 to 0.04], Standard Error of Mean 0.19

9. Secondary Outcome: Number of Participants With Treatment-Emergent Serious Adverse Events (SAEs)
Time Frame: Through day 29
Population: Safety Analysis Set (SAF): Randomized participants who received any study drug; based on the treatment received (as treated)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo IV Dose | 300mg IV | 600mg IV | 1200mg IV | 2400mg IV | Placebo SC Dose | 600mg SC | 1200mg SC
Number analyzed (Participants) | 82 | 165 | 162 | 165 | 166 | 82 | 163 | 164
Participants | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1

10. Secondary Outcome: Number of Participants With Infusion-Related Reactions Grade 2 or Above
Time Frame: Through day 4
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo IV Dose | 300mg IV | 600mg IV | 1200mg IV | 2400mg IV | Placebo SC Dose | 600mg SC | 1200mg SC
Number analyzed (Participants) | 82 | 165 | 162 | 165 | 166 | 82 | 163 | 164
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Injection-Site Reactions Grade 3 or Above
Time Frame: Through day 4
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo IV Dose | 300mg IV | 600mg IV | 1200mg IV | 2400mg IV | Placebo SC Dose | 600mg SC | 1200mg SC
Number analyzed (Participants) | 82 | 165 | 162 | 165 | 166 | 82 | 163 | 164
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Hypersensitivity Reactions Grade 2 or Above
Time Frame: Through day 29
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo IV Dose | 300mg IV | 600mg IV | 1200mg IV | 2400mg IV | Placebo SC Dose | 600mg SC | 1200mg SC
Number analyzed (Participants) | 82 | 165 | 162 | 165 | 166 | 82 | 163 | 164
Participants | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1

13. Secondary Outcome: Concentration of REGN10933 in Serum
Time Frame: Pre-Dose, 15 minutes Post-Dose, 3 days Post-Dose, 5 days Post-Dose, 7 days Post-Dose, 120 days Post-Dose
Population: Number Analyzed = number of participants contributing to each nominal timepoint
Measure: Mean (Standard Deviation); unit: milligrams per liter (mg/L)
Arm/Group | 300mg IV | 600mg IV | 1200mg IV | 2400mg IV | 600mg SC | 1200mg SC
Number analyzed (Participants) | 165 | 162 | 165 | 166 | 163 | 164
milligrams per liter (mg/L)
  Pre-dose: number analyzed (Participants) | 160 | 159 | 158 | 165 | 160 | 158
  Pre-dose | 0.529 (4.51) | 1.95 (12.1) | 0.847 (6.28) | 13.3 (130) | 0.992 (12.5) | 0.395 (4.96)
  15 minutes Post-Dose: number analyzed (Participants) | 162 | 157 | 161 | 163 | 158 | 157
  15 minutes Post-Dose | 58.2 (52.1) | 95.8 (57.9) | 178 (118) | 375 (267) | 8.73 (52.7) | 3.89 (19.7)
  3 days Post-Dose: number analyzed (Participants) | 162 | 155 | 156 | 164 | 158 | 155
  3 days Post-Dose | 32.5 (15.7) | 54.9 (19.2) | 109 (37.9) | 223 (63.9) | 22.4 (18.3) | 41.0 (19.3)
  5 days Post-Dose: number analyzed (Participants) | 158 | 152 | 160 | 162 | 154 | 160
  5 days Post-Dose | 27.7 (16.8) | 46.6 (16.9) | 88.4 (27.8) | 186 (53.3) | 26.3 (10.7) | 54.9 (34.0)
  7 days Post-Dose: number analyzed (Participants) | 159 | 157 | 161 | 161 | 159 | 160
  7 days Post-Dose | 23.9 (13.5) | 39.8 (11.5) | 82.8 (26.3) | 164 (46.0) | 26.8 (9.65) | 54.6 (19.9)
  120 days Post-Dose: number analyzed (Participants) | 152 | 139 | 150 | 149 | 148 | 141
  120 days Post-Dose | 1.78 (1.13) | 3.25 (1.88) | 6.46 (4.74) | 12.3 (8.42) | 2.73 (1.89) | 5.64 (3.77)

14. Secondary Outcome: Immunogenicity as Measured by Anti-drug Antibodies (ADAs) to REGN10933
Time Frame: Through day 120
Population: ADA analysis set includes all treated participants who received any amount of study drug and had at least one non-missing antibody variables result following the first dose of study drug or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo (IV + SC) | 300mg IV | 600mg IV | 1200mg IV | 2400mg IV | 600mg SC | 1200mg SC
Number analyzed (Participants) | 149 | 152 | 138 | 150 | 150 | 147 | 141
Participants
  Pre-existing Immunoreactivity | 3 | 2 | 3 | 0 | 2 | 1 | 3
  Treatment-Boosted Response | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Treatment-Emergent Response | 4 | 11 | 6 | 7 | 1 | 14 | 5
  Negative | 142 | 139 | 128 | 143 | 147 | 132 | 133

15. Secondary Outcome: Immunogenicity as Measured by Neutralizing Anti-drug Antibody (NAb) to REGN10933
Time Frame: Through day 120
Population: NAb analysis set includes all treated participants who received any study drug, had at least one non-missing antibody result following the first dose of study drug, and either tested negative at all ADA sampling times or tested positive for ADA with at least one non-missing NAb result after first dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo (IV + SC) | 300mg IV | 600mg IV | 1200mg IV | 2400mg IV | 600mg SC | 1200mg SC
Number analyzed (Participants) | 148 | 152 | 138 | 150 | 150 | 147 | 141
Participants
  Treatment-emergent & Treatment-boosted; Negative in NAb assay | 4 | 11 | 7 | 6 | 0 | 13 | 5
  Treatment-emergent & Treatment-boosted; Positive in NAb assay | 0 | 0 | 0 | 1 | 1 | 1 | 0
  ADA Negative | 142 | 139 | 128 | 143 | 147 | 132 | 133

16. Secondary Outcome: Concentration of REGN10987 in Serum
Time Frame: Pre-Dose, 15 minutes Post-Dose, 3 days Post-Dose, 5 days Post-Dose, 7 days Post-Dose, 120 days Post-Dose
Population: Number Analyzed = number of participants contributing to each nominal timepoint
Measure: Mean (Standard Deviation); unit: milligrams per liter (mg/L)
Arm/Group | 300mg IV | 600mg IV | 1200mg IV | 2400mg IV | 600mg SC | 1200mg SC
Number analyzed (Participants) | 165 | 162 | 165 | 166 | 163 | 164
milligrams per liter (mg/L)
  Pre-dose: number analyzed (Participants) | 160 | 159 | 158 | 165 | 160 | 158
  Pre-dose | 0.529 (4.38) | 2.04 (12.7) | 0.823 (6.48) | 13.1 (126) | 1.02 (12.8) | 0.370 (4.64)
  15 minutes Post-Dose: number analyzed (Participants) | 162 | 157 | 161 | 163 | 158 | 157
  15 minutes Post-Dose | 56.9 (53.1) | 95.4 (59.4) | 178 (119) | 383 (273) | 8.48 (51.7) | 4.36 (21.6)
  3 days Post-Dose: number analyzed (Participants) | 162 | 155 | 156 | 164 | 158 | 155
  3 days Post-Dose | 32.6 (15.9) | 56.0 (18.9) | 109 (38.5) | 225 (62.3) | 21.8 (16.2) | 42.0 (20.1)
  5 days Post-Dose: number analyzed (Participants) | 158 | 152 | 160 | 162 | 154 | 160
  5 days Post-Dose | 26.6 (15.5) | 46.3 (15.9) | 87.1 (26.9) | 177 (50.9) | 25.6 (9.31) | 52.9 (29.1)
  7 days Post-Dose: number analyzed (Participants) | 159 | 157 | 161 | 161 | 159 | 160
  7 days Post-Dose | 22.8 (12.8) | 38.0 (11.2) | 77.7 (24.3) | 151 (43.1) | 26.2 (8.74) | 53.7 (17.9)
  120 days Post-Dose: number analyzed (Participants) | 152 | 139 | 150 | 149 | 148 | 141
  120 days Post-Dose | 1.02 (0.805) | 1.97 (1.38) | 3.80 (3.10) | 6.88 (5.47) | 1.63 (1.43) | 3.26 (2.49)

17. Secondary Outcome: Immunogenicity as Measured by Anti-drug Antibodies (ADAs) to REGN10987
Time Frame: Through day 120
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo (IV + SC) | 300mg IV | 600mg IV | 1200mg IV | 2400mg IV | 600mg SC | 1200mg SC
Number analyzed (Participants) | 149 | 152 | 138 | 150 | 150 | 147 | 141
Participants
  Pre-existing Immunoreactivity | 3 | 4 | 0 | 3 | 3 | 3 | 3
  Treatment-Boosted Response | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Treatment-Emergent Response | 6 | 17 | 11 | 13 | 7 | 23 | 14
  Negative | 142 | 131 | 126 | 133 | 140 | 121 | 124

18. Secondary Outcome: Immunogenicity as Measured by Neutralizing Anti-drug Antibody (NAb) to REGN10987
Time Frame: Through day 120
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo (IV + SC) | 300mg IV | 600mg IV | 1200mg IV | 2400mg IV | 600mg SC | 1200mg SC
Number analyzed (Participants) | 148 | 152 | 138 | 150 | 150 | 147 | 141
Participants
  Pre-existing Immunoreactivity; Negative in NAb assay | 1 | 2 | 0 | 2 | 1 | 2 | 3
  Treatment-emergent & Treatment-boosted; Negative in NAb assay | 5 | 10 | 7 | 10 | 5 | 17 | 10
  Treatment-emergent & Treatment-boosted; Positive in NAb assay | 1 | 7 | 5 | 4 | 2 | 6 | 4
  ADA Negative | 140 | 131 | 126 | 133 | 140 | 121 | 124

ADVERSE EVENTS:
Time Frame: From first dose of study drug to Day 169
Groups:
- Placebo IV: Participants received a single intravenous dose of placebo matching REGN10933+REGN10987
- REGN10933 + REGN10987 300 mg IV: Participants received a single 300mg intravenous dose of REGN10933+REGN10987
- REGN10933 + REGN10987 600 mg IV: Participants received a single 600mg intravenous dose of REGN10933+REGN10987
- REGN10933 + REGN10987 1200 mg IV: Participants received a single 1200mg intravenous dose of REGN10933+REGN10987
- REGN10933 + REGN10987 2400 mg IV: Participants received a single 2400mg intravenous dose of REGN10933+REGN10987
- Placebo SC: Participants received a single subcutaneous dose of placebo matching REGN10933+REGN10987
- REGN10933 + REGN10987 600 mg SC: Participants received a single 600mg subcutaneous dose of REGN10933+REGN10987
- REGN10933 + REGN10987 1200 mg SC: Participants received a single 1200mg subcutaneous dose of REGN10933+REGN10987
Arm/Group | Placebo IV | REGN10933 + REGN10987 300 mg IV | REGN10933 + REGN10987 600 mg IV | REGN10933 + REGN10987 1200 mg IV | REGN10933 + REGN10987 2400 mg IV | Placebo SC | REGN10933 + REGN10987 600 mg SC | REGN10933 + REGN10987 1200 mg SC
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/165 | 0/162 | 0/165 | 0/166 | 0/82 | 0/163 | 0/164
Serious Adverse Events (participants affected / at risk) | 1/82 | 1/165 | 0/162 | 1/165 | 3/166 | 0/82 | 0/163 | 1/164
Other Adverse Events (participants affected / at risk) | 17/82 | 21/165 | 27/162 | 28/165 | 16/166 | 11/82 | 18/163 | 21/164
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo IV (N=82) | REGN10933 + REGN10987 300 mg IV (N=165) | REGN10933 + REGN10987 600 mg IV (N=162) | REGN10933 + REGN10987 1200 mg IV (N=165) | REGN10933 + REGN10987 2400 mg IV (N=166) | Placebo SC (N=82) | REGN10933 + REGN10987 600 mg SC (N=163) | REGN10933 + REGN10987 1200 mg SC (N=164)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary bladder rupture (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo IV (N=82) | REGN10933 + REGN10987 300 mg IV (N=165) | REGN10933 + REGN10987 600 mg IV (N=162) | REGN10933 + REGN10987 1200 mg IV (N=165) | REGN10933 + REGN10987 2400 mg IV (N=166) | Placebo SC (N=82) | REGN10933 + REGN10987 600 mg SC (N=163) | REGN10933 + REGN10987 1200 mg SC (N=164)
COVID-19 (Infections and infestations) | 17 (18) | 21 (21) | 27 (28) | 28 (29) | 16 (18) | 11 (11) | 18 (19) | 21 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/41/NCT04666441/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/41/NCT04666441/SAP_001.pdf